CLINICAL TRIAL: NCT06918054
Title: Hepatoprotective Measures for Children and Adolescents With Acute Lymphoblastic Leukemia During Induction Chemotherapy
Brief Title: Hepatoprotective for Children and Adolescent With Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU MD278/2023; FMASU MD278/2023 (Other: Faculty of Medicine Ain Shams University Research Ethical Committee)
Record Dates: First submitted 2024-12-06; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Leukaemia (Acute); Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Hepatoprotective program
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Implementation of a proposed whole program of monitoring and prevention of acute hepatic injury during the time of induction chemotherapy in children and adolescent with ALL.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Retrospective historical control (No Intervention): Retrospective historical control (Arm 1): Children and adolescent with ALL received Total XV induction chemotherapy from 1st June 2018 till 30th April 2023
- Interventional arm (Arm 2):Children and adolescent with ALL receiving Total XV induction chemotherap (Active Comparator): Implementation of hepatic supportive program
  1. Dietary modification: Patients will follow Mediterranean Diet (MD), this diet is characterized by a high intake of vegetables, fruit, whole cereals, legumes, nuts, and fish and a low intake of red meat and homemade desserts. The main added fat was extra virgin olive oil, with 35-40% kcal from fat (<10% from saturated fat), 40-44% kcal from carbohydrate, and 20% kcal from protein
  2. Evaluation of the risk of malnutrition in hospitalized children with cancer through SCAN score which is simple, quick and valid tool. A score of 0 - 1indicates a low risk of malnutrition. A score of 2 indicates a moderate risk of malnutrition. A score of 3 - 5 indicates a high risk of malnutrition.
  3. Supplementation of omega 3 fatty acids ( dose based on weight: <40 kg-450 mg/day, 40-60 kg-900 mg/day, >60 kg-1300 mg/day)
  Interventions: Dietary Supplement: Dietary modification; Dietary Supplement: Supplementation of omega 3 fatty acids

INTERVENTIONS:
Dietary Supplement: Dietary modification — Patients will follow Mediterranean Diet (MD), this diet is characterized by a high intake of vegetables, fruit, whole cereals, legumes, nuts, and fish and a low intake of red meat and homemade desserts. The main added fat was extra virgin olive oil, with 35-40% kcal from fat (<10% from saturated fat), 40-44% kcal from carbohydrate, and 20% kcal from protein
  Arms: Interventional arm (Arm 2):Children and adolescent with ALL receiving Total XV induction chemotherap
Dietary Supplement: Supplementation of omega 3 fatty acids — Supplementation of omega 3 fatty acids ( dose based on weight: <40 kg-450 mg/day, 40-60 kg-900 mg/day, >60 kg-1300 mg/day)
  Arms: Interventional arm (Arm 2):Children and adolescent with ALL receiving Total XV induction chemotherap

SUMMARY:
This current study will implement a proposed whole program of monitoring and prevention acute hepatic injury during the time of induction chemotherapy in children and adolescent with ALL.

DETAILED DESCRIPTION:
Children and adolescent with acute lymphoblastic leukemia (ALL) can exhibit a wide spectrum of hepatotoxicity ranging from asymptomatic to clinically significant during induction chemotherapy. Unmonitored hepatic status can lead to a hepatic toxicity that might result in unwarranted interruption of the aimed delivery of dose dense chemotherapy to induce remission and consequent treatment.

To evaluate the effect of chemotherapy in children and adolescent with ALL during induction phase, through recording liver function tests before, during and after induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Children and adolescents aged from 2 to 18 years newly diagnosed with acute lymphoblastic leukemia during induction phase of chemotherapy treated at Ain Shams

Exclusion Criteria:

Known chronic liver disease.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Implementation a program of hepatic support | Almost 1 year
  To implement a hepatoprotection interventional program to children and adolescent with ALL during Total XV induction c

CONTACTS AND LOCATIONS:
Overall Officials: Manal El-Sayed, MD, Study Chair — Faculty of Medicine Ain Shams University
Locations (2):
- Egypt (2):
  - Ain Shams University, Cairo
  - Faculty of Medicine Ain Shams Research Institute- Clinical Research Center (MASRI-CRC), Cairo